CLINICAL TRIAL: NCT01115322
Title: A Phase 1, Evaluator-Blinded, Randomized, Vehicle Controlled Study To Evaluate The Phototoxic Potential Of Topically Applied Tazarotene Foam In Healthy Volunteers
Brief Title: A Study to Evaluate the Potential of Tazarotene Foam to Cause a Reaction When Applied to the Skin and Exposed to Light on Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 114573
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Acne Vulgaris
Keywords: Healthy volunteer study; phototoxicity
MeSH Terms: conditions — Acne Vulgaris; Dermatitis, Phototoxic | interventions — Radiation; Light

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Tazarotene Foam without irradiation (Experimental): Subjects will be exposed to Tazarotene Foam Patch without irradiation
  Interventions: Drug: Tazarotene Foam without irradiation
- Tazarotene Foam with UVA and UVB irradiation (Experimental): Subjects will be exposed to Tazarotene Foam Patch with UVA and UVB irradiation
  Interventions: Drug: Tazarotene Foam with UVA and UVB irradiation
- Tazarotene Foam with UVA , UVB, and visible light irradiation (Experimental): Subjects will be exposed to Tazarotene Foam with UVA and UVB and visible light irradiation
  Interventions: Drug: Tazarotene Foam with UVA, UVB, and visible light
- Vehicle Foam without irradiation (Placebo Comparator): Subjects will be exposed to Vehicle Foam Patch without irradiation
  Interventions: Drug: Vehicle Foam without irradiation
- Vehicle Foam with UVA and UVB irradiation (Placebo Comparator): Subjects will be exposed to Vehicle Foam Patch with UVA and UVB irradiation
  Interventions: Drug: Vehicle Foam with UVA and UVB irradiation
- Vehicle Foam with UVA and UVB and visible light irradiation (Placebo Comparator): Subjects will be exposed to Vehicle Foam Patch with UVA and UVB and visible light irradiation
  Interventions: Drug: Vehicle Foam with UVA and UVB and visible light irradiation
- No Treatment without irradiation (Sham Comparator): Subjects will be exposed to a Blank Patch without irradiation
  Interventions: Drug: No Treatment without irradiation
- No Treatment with UVA and UVB irradiation (Sham Comparator): Subjects will be exposed to a Blank Patch with UVA and UVB irradiation
  Interventions: Drug: No Treatment with UVA and UVB irradiation
- No Treatment with UVA and UVB and visible light irradiation (Sham Comparator): Subjects will be exposed to a Blank Patch with UVA and UVB and visible light irradiation
  Interventions: Drug: No Treatment with UVA and UVB and visible light irradiation

INTERVENTIONS:
Drug: Tazarotene Foam without irradiation — Each subject will be exposed to a patch with tazarotene foam during a single, 24 hour application period.
  This patch will then be removed and those sites will serve as nonirradiated control. Patch sites will be evaluated for signs of inflammatory skin responses (eg, erythema and local skin reactions) and superficial effects 1 ±0.25 hour after patch removal, and during follow-up visits at 24 ±1 hours, 48 ±2 hours, and 72 ±2 hours after patch removal.
  Arms: Tazarotene Foam without irradiation
Drug: Tazarotene Foam with UVA and UVB irradiation — Each subject will be exposed to a patch with tazarotene foam during a single, 24 hour application period. The patch will be removed and that site will be exposed to ultraviolet A (UVA) and to UVA/ultraviolet B (UVB) radiation wavelengths (UV only).
  Patch sites will be evaluated for signs of inflammatory skin responses (eg, erythema and local skin reactions) and superficial effects 1 ±0.25 hour after patch removal, and during follow-up visits at 24 ±1 hours, 48 ±2 hours, and 72 ±2 hours after patch removal.
  Arms: Tazarotene Foam with UVA and UVB irradiation
Drug: Tazarotene Foam with UVA, UVB, and visible light — Each subject will be exposed to a patch with tazarotene foam during a single, 24 hour application period. The patch will be removed and that site will be exposed to UVA, UVA/UVB, and visible light (VIS) wavelengths (UV plus VIS).
  Patch sites will be evaluated for signs of inflammatory skin responses (eg, erythema and local skin reactions) and superficial effects 1 ±0.25 hour after patch removal, and during follow-up visits at 24 ±1 hours, 48 ±2 hours, and 72 ±2 hours after patch removal.
  Arms: Tazarotene Foam with UVA , UVB, and visible light irradiation
Drug: Vehicle Foam without irradiation — Each subject will be exposed to a patch with vehicle foam during a single, 24 hour application period. This patch will then be removed and those sites will serve as nonirradiated control. Patch sites will be evaluated for signs of inflammatory skin responses (eg, erythema and local skin reactions) and superficial effects 1 ±0.25 hour after patch removal, and during follow-up visits at 24 ±1 hours, 48 ±2 hours, and 72 ±2 hours after patch removal.
  Arms: Vehicle Foam without irradiation
Drug: Vehicle Foam with UVA and UVB irradiation — Each subject will be exposed to a patch with vehicle foam during a single, 24 hour application period. The patch will be removed and that site will be exposed to ultraviolet A (UVA) and to UVA/ultraviolet B (UVB) radiation wavelengths (UV only).
  Patch sites will be evaluated for signs of inflammatory skin responses (eg, erythema and local skin reactions) and superficial effects 1 ±0.25 hour after patch removal, and during follow-up visits at 24 ±1 hours, 48 ±2 hours, and 72 ±2 hours after patch removal.
  Arms: Vehicle Foam with UVA and UVB irradiation
Drug: Vehicle Foam with UVA and UVB and visible light irradiation — Each subject will be exposed to a patch with vehicle foam during a single, 24 hour application period. The patch will be removed and that site will be exposed to UVA, UVA/UVB, and visible light (VIS) wavelengths (UV plus VIS).
  Patch sites will be evaluated for signs of inflammatory skin responses (eg, erythema and local skin reactions) and superficial effects 1 ±0.25 hour after patch removal, and during follow-up visits at 24 ±1 hours, 48 ±2 hours, and 72 ±2 hours after patch removal.
  Arms: Vehicle Foam with UVA and UVB and visible light irradiation
Drug: No Treatment without irradiation — Each subject will be exposed to a blank patch during a single, 24 hour application period. This patch will then be removed and those sites will serve as nonirradiated control. Patch sites will be evaluated for signs of inflammatory skin responses (eg, erythema and local skin reactions) and superficial effects 1 ±0.25 hour after patch removal, and during follow-up visits at 24 ±1 hours, 48 ±2 hours, and 72 ±2 hours after patch removal.
  Arms: No Treatment without irradiation
Drug: No Treatment with UVA and UVB irradiation — Each subject will be exposed to a blank patch during a single, 24 hour application period. The patch will be removed and that site will be exposed to ultraviolet A (UVA) and to UVA/ultraviolet B (UVB) radiation wavelengths (UV only).
  Patch sites will be evaluated for signs of inflammatory skin responses (eg, erythema and local skin reactions) and superficial effects 1 ±0.25 hour after patch removal, and during follow-up visits at 24 ±1 hours, 48 ±2 hours, and 72 ±2 hours after patch removal.
  Arms: No Treatment with UVA and UVB irradiation
Drug: No Treatment with UVA and UVB and visible light irradiation — Each subject will be exposed to a blank patch during a single, 24 hour application period. The patch will be removed and that site will be exposed to UVA, UVA/UVB, and visible light (VIS) wavelengths (UV plus VIS).
  Patch sites will be evaluated for signs of inflammatory skin responses (eg, erythema and local skin reactions) and superficial effects 1 ±0.25 hour after patch removal, and during follow-up visits at 24 ±1 hours, 48 ±2 hours, and 72 ±2 hours after patch removal.
  Arms: No Treatment with UVA and UVB and visible light irradiation

SUMMARY:
The purpose of this study is to evaluate the potential of Tazarotene Foam to induce a phototoxic reaction when exposed to UV and VIS light on skin of healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, single center, evaluator-blinded, randomized, vehicle controlled study to evaluate the potential of Tazarotene Foam 0.1% to induce a phototoxic reaction in healthy adult volunteers. Approximately 40 healthy, male and female, volunteer subjects aged 18 to 65 years will be enrolled.

Each subject will be exposed to three (3) sets of three (3) patches containing Tazarotene Foam, Vehicle Foam and a Blank Patch (no study product). Each patch set will be applied to randomized sites on the subject's back. Patch sets will be removed and evaluated after 24 hours of exposure. The exposed patch sites will then be irradiated (exposed to light) and evaluated at 1 hour post irradiation and at 24, 48, and 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed and dated written voluntary informed consent and Health Information Portability and Accountability Act (HIPAA) authorization before any protocol-specific procedures are performed.
* Male or female aged 18 to 65 years, inclusive, at time of consent.
* Able and willing to complete the study and to comply with all study instructions.
* Possess Fitzpatrick skin types I (always burns easily; never tans), II (always burns easily; tans minimally), or III (burns moderately; tans gradually) that will not interfere with the evaluation of any skin responses (Fitzpatrick 1988). Determination of skin types will be based on sunburn and tanning histories, as well as subjects' opinions of their responses to the first 30 to 45 minutes of sun exposure.
* Male subjects and their partners must agree to use a medically acceptable method of contraception.

Additional criteria for women of childbearing potential, defined as one who is biologically capable of becoming pregnant, including perimenopausal women who are less than 2 years from their last menses:

* A regular menstrual cycle before study entry (as reported by the subject).
* Negative urine pregnancy test within 2 weeks of the first application of study product.
* Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception throughout the duration of the study. Acceptable contraceptive methods include the following:

  * Hormonal contraception, including oral, injectable, or implantable methods started at least 2 months prior to screening. If hormonal contraception was started less than 2 months prior to screening, then a form of nonhormonal contraception should be added until the third continuous month of hormonal contraception has been completed.
  * Two forms of reliable nonhormonal contraception, to include the use of either an intrauterine device plus a reliable barrier method or 2 reliable barrier methods. Reliable barrier methods include condoms or diaphragms. A cervical cap is also a reliable barrier method, provided that the female subject has never given birth vaginally. The combined use of a condom and spermicide constitute 2 forms of acceptable nonhormonal contraception, provided that they are both used properly. The use of spermicide alone and the improper use of condoms are inferior methods of contraception. Subjects with surgical sterilization, including tubal sterilization or partner's vasectomy, must use a form of nonhormonal contraception. A barrier method or sterilization plus spermicide is acceptable.

Women who are not currently sexually active must agree to use a medically acceptable method of contraception should they become sexually active while participating in the study.

Exclusion Criteria:

* Female who is pregnant, trying to become pregnant, or breast feeding.
* Considered unable or unlikely to attend the necessary visits.
* History of known or suspected intolerance to tazarotene, any of the ingredients of the study products, the hypoallergenic tape, or the cotton patches.
* Participation in any patch test study within 4 weeks of Screening Visit 1.
* Inability to evaluate the skin in and around the potential patch test sites on the back due to sunburns, unevenness in skin tones, tattoos, scars, excessive hair, freckles, birthmarks, moles, or other skin damage or abnormality.
* Clinically significant skin diseases that may contraindicate participation or interfere with patch test site evaluations, including psoriasis, eczema, atopic dermatitis, acne, dysplastic nevi, or other skin pathologies, or a history of skin cancer.
* A history of severe reactions from exposure to sunlight, including previous experience with photoallergy, solar urticaria, polymorphous light eruptions, or other photo exacerbated systemic diseases.
* Any major illness within 4 weeks of Screening Visit 1.
* Considered immunocompromised.
* A clinically relevant history of or current evidence of abuse of alcohol or other drugs.
* Clinically relevant history or currently suffering from any disease or condition that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk. This may include respiratory (including chronic asthma requiring repetitive drug interventions), gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, or connective tissue diseases or disorders.
* Used photosensitizing medications (prescription, nonprescription, or herbal) or a known photosensitizing material within 2 weeks of Screening Visit 1.
* Received any investigational product or procedure within 4 weeks of Screening Visit 1 or is scheduled to receive an investigational product (other than the study product) or procedure during the study.
* Received allergy injections within 1 week of Screening Visit 1, or expects to receive allergy injections during study participation.
* Received immunizations within 4 weeks of Screening Visit 1.
* Used systemic or topical corticosteroids or other immunosuppressive medications within 4 weeks of Screening Visit 1.
* Used topical medications or other products (eg, self tanning products, waxing products, benzoyl peroxide, salicylic acid, or sulfur) in the areas of patch testing within 2 weeks of Screening Visit 1.
* Used antihistamines, selective leukotriene receptor antagonists (eg, montelukast sodium, zafirlukast), or mast cell stabilizers (eg, cromolyn sodium or nedocromil sodium) within 4 weeks of Screening Visit 1.
* Used nonsteroidal anti inflammatory medications within 2 weeks of Screening Visit 1.
* Currently using any medication that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
* Participated in a previous study of the same study product.
* Employee of the study center, contract research organization, or Stiefel who is involved in the study, or an immediate family member (eg, partner, offspring, parents, siblings or sibling's offspring) of an employee who is involved in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2010-04-10 (Actual); Study Completion 2010-04-10 (Actual)

PRIMARY OUTCOMES:
Inflammatory skin responses | Day 2-5 (24, 48, 72 hours following patch application).
  Evaluation of patch sites for inflammatory skin responses and superficial effects following 24 hours of exposure and following irradiation on Day 2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- HillTop Research Corporation, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Hogan DJ, Saenz AB. Phototoxic and photoallergic potential of tazarotene foam 0.1% in 2 phase 1 patch studies. Cutis. 2012 Nov;90(5):266-71. PMID 23270200
- See also: Results for study 114573 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114573?search=study&search_terms=114573#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 114573 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114573 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114573 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114573 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114573 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114573 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114573 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register